CLINICAL TRIAL: NCT02667002
Title: Randomized Single Blind Controlled Trial of Comparison of Anatomic and Sexual Outcomes Between Conventional and Bilateral Sacral Hysteropexy
Brief Title: Comparison of Anatomic Results Between Bilateral and Conventional Abdominal Sacral Hysteropexy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeynep Kamil Maternity and Pediatric Research and Training Hospital (Other)
Responsible Party: Principal Investigator, Mehmet Baki Senturk, Principal Investigator, Zeynep Kamil Maternity and Pediatric Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 162
Record Dates: First submitted 2016-01-21; First posted 2016-01-28 (Estimated); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Bilateral Abdominal Sacral Hysteropexy (Experimental): Bilateral abdominal sacral hysteropexy will be perform in 10 patients. One month after patients will be evaluate by MRI and Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12) form.
  Interventions: Procedure: Bilateral Abdominal Sacral Hysteropexy
- Classic Abdominal Sacral Hysteropexy (Experimental): Conventional abdominal sacral hysteropexy will be perform in 10 patients. One month after patients will be evaluate by MRI and Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12) form.
  Interventions: Procedure: Conventional abdominal Sacral Hysteropexy
- Women with no uterovaginal prolapsed (Active Comparator): Ten nulliparous participants with no uterovaginal prolapsed will be evaluate by MRI and Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12) form.
  Interventions: Other: Nulliparous women with no uterovaginal prolapsed

INTERVENTIONS:
Procedure: Bilateral Abdominal Sacral Hysteropexy — The mesh will be fixed right and left side of sacrum.
  Arms: Bilateral Abdominal Sacral Hysteropexy
Procedure: Conventional abdominal Sacral Hysteropexy — The mesh will be fixed only right side of sacrum
  Arms: Classic Abdominal Sacral Hysteropexy
Other: Nulliparous women with no uterovaginal prolapsed — This will be control group which consistent patients with no uterovaginal prolapse.
  Arms: Women with no uterovaginal prolapsed

SUMMARY:
Investigators separated 20 patients with uterovaginal prolapse into 2 groups according to random numbers table. In one group, conventional abdominal sacral hysteropexy will be perform and another group bilateral abdominal sacral hysteropexy will be perform with polypropylene mesh. After 1 mont operation vaginal configuration will be evaluate with MRI on three plane (axial, sagittal, coronal). Then the results of thus two groups will be compare to results of nullipara patients. Investigators will investigate which technique keep the vaginal axis is closer to the original anatomic position.

DETAILED DESCRIPTION:
Since vaginal hysterectomy and mc call culdoplasty, many techniques have been described. Before, correcting only prolapsed part, now, we can measure anatomical and functional results more objectively by using different tool such us MRI, perineal ultrasonography, PISQ-12, IIQ-7 (Incontinence impact questionnaire). Hence pelvic organ prolapse surgery is important in terms of anatomic and functional results. Unilateral abdominal sacral hysteropexy can put vaginal axis to right side slightly. Therefore investigators hypothesized that bilateral sacral hysteropexy which mimic sacrouterine ligament can be more suitable in terms of anatomic results.

ELIGIBILITY:
Inclusion Criteria:

* Women with stage 3 or more pelvic organ prolapse

Exclusion Criteria:

* Women with abnormal uterine bleeding, abnormal cervical screening test, myoma uteri and want to hysterectomy

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-05 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Anatomic Success | One month
  anatomic success will be evaluated by using magnetic resonance imaging. Vaginal axis (distance to spin ischiadic a and sacrum) will be measure on three plane

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Baki Şentürk, MD, Study Director — Zeynep Kamil Maternity and Pediatric Research and Training Hospital

IPD SHARING:
Plan to Share IPD: Yes
Data will be available within 1 week of study completion.

REFERENCES:
- [Result] Jager W, Mirenska O, Brugge S. Surgical treatment of mixed and urge urinary incontinence in women. Gynecol Obstet Invest. 2012;74(2):157-64. doi: 10.1159/000339972. Epub 2012 Aug 9. PMID 22890409
- [Result] Sze EH, Meranus J, Kohli N, Miklos JR, Karram MM. Vaginal configuration on MRI after abdominal sacrocolpopexy and sacrospinous ligament suspension. Int Urogynecol J Pelvic Floor Dysfunct. 2001;12(6):375-9; discussion 379-80. doi: 10.1007/s001920170016. PMID 11795640
- [Result] Joukhadar R, Meyberg-Solomayer G, Hamza A, Radosa J, Bader W, Barski D, Ismaeel F, Schneider G, Solomayer E, Baum S. A Novel Operative Procedure for Pelvic Organ Prolapse Utilizing a MRI-Visible Mesh Implant: Safety and Outcome of Modified Laparoscopic Bilateral Sacropexy. Biomed Res Int. 2015;2015:860784. doi: 10.1155/2015/860784. Epub 2015 Apr 19. PMID 25961042
- See also: pubmed — http://www.ncbi.nlm.nih.gov/pubmed/22890409
- See also: pubmed — http://www.ncbi.nlm.nih.gov/pubmed/25961042
- See also: pubmed — http://www.ncbi.nlm.nih.gov/pubmed/?term=Vaginal+Configuration+on+MRI+after+Abdominal+Sacrocolpopexy+and+Sacrospinous+Ligament+Suspension